CLINICAL TRIAL: NCT04255420
Title: Sphenopalatine Ganglion Blocks for Headaches in the Emergency Department
Brief Title: SPG Blocks for Headaches
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kendall Healthcare Group, Ltd. (Industry)
Collaborators: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSU IRB 2019-48
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Headache
Keywords: sphenopalatine ganglion block
MeSH Terms: conditions — Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SPG Block (Experimental): Sphenopalatine ganglion block using cotton-tipped applicators soaked in 1% lidocaine will be performed.
  Interventions: Procedure: SPG Block
- Standard Treatment (Active Comparator): Intravenous prochlorperazine 10 mg plus diphenhydramine 50 mg.
  Interventions: Drug: Standard IV Treatment

INTERVENTIONS:
Procedure: SPG Block — A cotton-tipped applicator soaked in 1% lidocaine will be inserted into the nostril on the side of the headache. If the headache is bilateral, two cotton-tipped applicators will be inserted. The cotton-tipped applicators will be left in place for 15 minutes.
  Arms: SPG Block
Drug: Standard IV Treatment — Intravenous prochlorperazine 10 mg plus diphenhydramine 50 mg will be administered.
  Arms: Standard Treatment

SUMMARY:
This will be a single-center, open-label clinical trial comparing sphenopalatine ganglion blocks to standard intravenous therapy for patients who come to the emergency department for a headache.

DETAILED DESCRIPTION:
Having outperformed other agents in head-to-head trials, intravenous (IV) dopamine antagonists, such as prochlorperazine or metoclopramide, are generally considered the 1st line treatment for headaches in the ED. However, despite the relative effectiveness of prochlorperazine, a substantial number of patients who present to the ED with a headache still have a moderate to severe headache 24 hours after discharge. Moreover, some patients may have difficult IV access, so it would be useful to employ a technique that could effectively treat headaches without the use of an IV line.

One therapy that has been suggested but not well-studied that might help treat headaches in the ED without the use of an IV line is the sphenopalatine ganglion (SPG) block via intranasal lidocaine. The sphenopalatine ganglion may play a role in the development of pain in primary headaches through the release of neuropeptides that activate or sensitize intracranial nociceptors. Several prior randomized trials have evaluated the use of intranasal lidocaine or bupivacaine vs placebo for patients with migraine headaches, and the results have been mixed.

Thus, the investigators propose a single-center, open-label, clinical trial to compare the efficacy of SPG blocks to standard IV therapy for headaches in the ED.

Adult patients who come to the ED for a suspected primary headache may be enrolled. Patients who are assigned to the standard IV therapy group will receive prochlorperazine 10 mg and diphenhydramine 50 mg.

Patients who are assigned to the SPG block group will undergo the following procedure. A cotton-tipped applicator soaked in 1% lidocaine will be placed in the nostril on the side of the headache. If the headache is bilateral, a cotton-tipped applicator will be inserted into each nostril. The cotton-tipped applicator(s) will be left in place for 15 minutes. If the patient has not had significant improvement upon removal of the cotton-tipped applicator the physician may order IV medication for the patient's headache ("rescue analgesia").

Just before the initiation of treatment, an initial visual analog scale (VAS) pain score will be obtained from the patient. The VAS pain score will be repeated 15 and 30 minutes after treatment. Additional data will be determined through chart review and telephone follow up with the patient 24-72 hours after discharge.

The primary outcome of the study will be the difference between groups in the fraction of patients with a 50% reduction in VAS pain score at 15 minutes. Secondarily, the investigators will compare groups with regards to their mean VAS pain scores as 15 and 30 minutes after the initiation of the first treatment, hospital length of stay, the need for rescue analgesic medications, complications (nose bleed, akathisia, etc.), and presence of persistent headache 24-72 hours after discharge on telephone follow up.

ELIGIBILITY:
Inclusion Criteria:

* Any patient at least 18 years old who presented to the ED with a suspected primary headache.

Exclusion Criteria:

* pregnant women
* prisoners
* meningeal signs
* fever
* any acute abnormality on neurologic exam
* allergy to one of study drugs
* on oral anticoagulant
* already received analgesic treatment in the ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients with Substantial Pain Reduction at 15 minutes | 15 minutes
  The percentage of patients whose 100 mm visual analog scale pain score reduced by at least 50% from before treatment until 15 minutes after the start of treatment.

SECONDARY OUTCOMES:
Change in Mean Pain Score at 15 minutes | 15 minutes
  The difference in the mean 100 mm visual analog scale pain score from before treatment to 15 minutes after treatment, and the means for each group will be compared.
Change in Mean Pain Score at 30 minutes | 30 minutes
  The difference in the mean 100 mm visual analog scale pain score from before treatment to 15 minutes after treatment, and the means for each group will be compared.
Headache 24-72 hours later | 24-72 hours
  Patients will be called by phone 24-72 hours after treatment in the ED to ask if they are having a headache (yes or no). The percentage of patients with a headache at that time will be compared between the groups.
Hospital Length of Stay | 30 minutes to 1 week
  The mean length of time the patient remains in the hospital will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Zitek, MD, Principal Investigator — Kendall Healthcare Group, Ltd.
Locations (1):
- Kendall Regional Medical Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: After completion of data analysis, the data will be available indefinitely.

REFERENCES:
- [Result] Yarnitsky D, Goor-Aryeh I, Bajwa ZH, Ransil BI, Cutrer FM, Sottile A, Burstein R. 2003 Wolff Award: Possible parasympathetic contributions to peripheral and central sensitization during migraine. Headache. 2003 Jul-Aug;43(7):704-14. doi: 10.1046/j.1526-4610.2003.03127.x. PMID 12890124
- [Result] Maizels M, Geiger AM. Intranasal lidocaine for migraine: a randomized trial and open-label follow-up. Headache. 1999 Sep;39(8):543-51. doi: 10.1046/j.1526-4610.1999.3908543.x. PMID 11279969
- [Result] Blanda M, Rench T, Gerson LW, Weigand JV. Intranasal lidocaine for the treatment of migraine headache: a randomized, controlled trial. Acad Emerg Med. 2001 Apr;8(4):337-42. doi: 10.1111/j.1553-2712.2001.tb02111.x. PMID 11282668
- [Result] Mohammadkarimi N, Jafari M, Mellat A, Kazemi E, Shirali A. Evaluation of efficacy of intra-nasal lidocaine for headache relief in patients refer to emergency department. J Res Med Sci. 2014 Apr;19(4):331-5. PMID 25097606
- [Result] Avcu N, Dogan NO, Pekdemir M, Yaka E, Yilmaz S, Alyesil C, Akalin LE. Intranasal Lidocaine in Acute Treatment of Migraine: A Randomized Controlled Trial. Ann Emerg Med. 2017 Jun;69(6):743-751. doi: 10.1016/j.annemergmed.2016.09.031. Epub 2016 Nov 23. PMID 27889366
- [Result] Schaffer JT, Hunter BR, Ball KM, Weaver CS. Noninvasive sphenopalatine ganglion block for acute headache in the emergency department: a randomized placebo-controlled trial. Ann Emerg Med. 2015 May;65(5):503-10. doi: 10.1016/j.annemergmed.2014.12.012. Epub 2015 Jan 7. PMID 25577713
- [Result] Maizels M, Scott B, Cohen W, Chen W. Intranasal lidocaine for treatment of migraine: a randomized, double-blind, controlled trial. JAMA. 1996 Jul 24-31;276(4):319-21. PMID 8656545